CLINICAL TRIAL: NCT06326944
Title: Analgesic Effect of Fascia Transversalis Block Versus Transversus Abdominal Plane Block in Children Undergoing Open Inguinal Hernia Surgery. A Randomized Comparative Trial.
Brief Title: Fascia Transversalis Versus Transversus Abdominis Plane Block for Children Undergoing Inguinal Hernia Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, maged gamal, Anesthesia lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-527-2023
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Fascia Transversalis Plane Block
Keywords: Transversus abdominis plane block; Open inguinal herniorrhaphy
MeSH Terms: interventions — Fentanyl; Meperidine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive fascia transversalis block
  Interventions: Procedure: Ultrasound- guided Fascia Transversalis plane block; Drug: Fentanyl; Drug: Pethidine; Drug: Acetaminophen
- Group B (Active Comparator): Patients will receive Transversus abdominus plane block
  Interventions: Procedure: Ultrasound-guided Transversus abdominus plane block; Drug: Fentanyl; Drug: Pethidine; Drug: Acetaminophen

INTERVENTIONS:
Procedure: Ultrasound- guided Fascia Transversalis plane block — Ultrasound probe will be placed in a transverse orientation above the iliac crest; and the external oblique, internal oblique (IO), and transversus abdominis TA muscles will be identified and traced posteriorly until first the TA muscle and then the IO muscle tapered into their common aponeurosis, adjacent to the quadratus lumborum muscle. The tip of a 22-gauge 80-mm block needle will be positioned just deep to the TA muscle and its aponeurosis at the point where the TA is tapered off. 0.4 ml/kg bupivacaine 0.25% will be injected into the plane between the TA and underlying transversalis fascia
  Arms: Group A
Procedure: Ultrasound-guided Transversus abdominus plane block — the probe will be placed transversely in the mid-axillary line between the iliac crest and the costal margin at the level of the umbilicus. The external oblique, internal oblique and transversus abdominis muscles and their fascias will be visualized. A 22 gauge, 80 mm needle will be introduced anteriorly and in the plane of the ultrasound probe, and on entering the plane between IO and TA, 2 ml of 0.9% saline will be injected to verify the correct position of the needle. Following negative aspiration, 0.4 ml/kg of bupivacaine 0.25% will be injected.
  Arms: Group B
Drug: Fentanyl — patients will receive an induction dose at 1 mcg/kg. If the analgesia was inadequate in the form of increase in heart rate and or arterial blood pressure by more than 20% of baseline values during surgery, this warrants the administration of intravenous fentanyl (0.5µg/kg).
Drug: Pethidine — Pethidine IV will be given as rescue analgesia (0.5 mg/kg) if the FLACC pain score was more than 4 , the maximum allowed dose is 1mg/kg every 4 hours.
  Other Names: Rescue analgesia
Drug: Acetaminophen — patients will be given paracetamol (15 mg /kg/8 hrs ).

SUMMARY:
Fascia transversalis block in pediatrics undergoing inguinal surgical repair may be simple technique and may give longer effect in reduction of post-operative pain in comparison to transversus abdominis plane block.

DETAILED DESCRIPTION:
All children will be assessed clinically, and investigations will be done to exclude the exclusion criteria mentioned above. Laboratory works needed: complete blood count (CBC), prothrombin time, concentration, partial thromboplastin time Intra-operative management Premedication by intramuscular injection of atropine 0.02 mg/Kg and midazolam 0.2 mg/Kg will be followed by insertion of intravenous (I.V) cannula.

General anesthesia will be induced in supine position under standard basic monitoring of vital signs with inhalational anesthetic using (100%) O2 + Sevoflurane. After deepening of the anesthesia, atracurium 0.5mg/kg and fentanyl 1μg/kg patients will be given, Endotracheal intubation will then follow by appropriate size of endotracheal tube. Volume control ventilation (VCV) 5-7 ml/kg and respiratory rate will be adjusted to keep and PaCO2 levels between 30-35 mmHg using (G.E-Datex-Ohmeda, Avance CS2, USA) anesthesia machine. Anesthesia will be maintained with isoflurane 1 MAC with 50% oxygen in air, and atracurium top-ups of 0.1mg/kg will be given every 30 minutes for neuromuscular blockade.

The Block will be performed using Sonosite S-Nerve Portable Ultrasound and SLAX/13-6 MHZ transducer will be used. 0.4 ml/kg bupivacaine 0.25% will be installed in the block plane. After receiving the block, surgical incision will be allowed to be done after 15 minutes.

Continuous recording of heart rate, blood pressure, will be carried out from the moment of injection at timely intervals intra-operative.

Increase of HR BP. >30% of baseline Indicates failure of block so fentanyl will be given at 1 mic / kg intra-operative.

Postoperative pain assessment using FLACC score will then follow till 6 hours

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II

Exclusion Criteria:

* Parents' refusal to participate in the study.
* Coagulopathy (i.e. Platelets ≤ 50,000 and/or INR> 1.5).
* Localized infection at the site of needle insertion.
* Known hypersensitivity or allergies to any of the used drugs.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Time to First need of analgesia | First 6 hours postoperative
  time (minutes) to First need of rescue analgesia

SECONDARY OUTCOMES:
Total Pethidine Consumption | First 6 hours postoperative
  Total postoperative rescue morphine consumption in mg/kg for each group in the first 24 hours post-operative period.
Postoperative pain assessment FLACC | First 6 hours postoperative
  In the PACU, quality of analgesia was assessed every 15 minutes for the first hour then at 2,4 ,and 6 hours postoperative using (face, legs, activity, and cry consolability scale) (FLACC) pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided